CLINICAL TRIAL: NCT06647147
Title: Impact of Aerobic Training on Lung Function in Women With Fibromyalgia
Brief Title: Aerobic Training on Lung Function in Fibromyalgia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Middle East University (Other)
Responsible Party: Principal Investigator, Saher Lotfy El Gayar, Assistant Professor of Physiotherapy, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Aerobic Training
Record Dates: First submitted 2024-10-16; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Fibromyalgia (FM); Respiration Disorders
MeSH Terms: conditions — Fibromyalgia; Respiration Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Active Comparator): 40 women with fibromyalgia will participate in low to moderate intensity aerobic training plus diaphragmatic breathing exercises.
  Interventions: Other: Aerobic training; Other: Diaphragmatic breathing exercises
- Control group (Active Comparator): 40 women with fibromyalgia will only participate in diaphragmatic breathing exercises.
  Interventions: Other: Diaphragmatic breathing exercises

INTERVENTIONS:
Other: Aerobic training — For twelve weeks, the women in the study group will participate in aerobic training on cycle ergometer. Each session will consist of 30-45 minutes of cycling at a moderate intensity, accompanied by a workout heart rate ranging from 65% to 75% of the maximal heart rate and ranging between 12 and 14 on the Borg rating of perceived exertion 20-point scale. After ten minutes of warm-up, every session will end with a brief 3-minute period of cool-down.
  Arms: Study group
Other: Diaphragmatic breathing exercises — From the hook-lying position, the women will receive instructions to position their hands on the rectus abdominis muscle located under the anterior chest wall. They will be advised to inhale slowly and deeply, expanding their abdomen without causing any movement in their upper chest, while simultaneously relaxing their shoulders. Slowly, the women will expel every breath. Air will be inhaled via the nose, swelling the abdomen. After the breath ceased, the women will purse her lips and exhale from his mouth with half-opened lips and a hollow belly. A single respiratory cycle consists of a three-second intake, followed by a three-second pause, and concluding with a six-second expiration phase.

SUMMARY:
Exploring the effect of aerobic exercises on lung function, chest movement, and exercise capacity in women suffering from fibromyalgia.

DETAILED DESCRIPTION:
Eighty women with fibromyalgia will be equally randomly assigned to the experimental (EX) group and the control group (CON). The participants' age will be between 30 and 40 years and they will have mild restrictive lung affection. The Ex group will attend 3 sessions/week of aerobic training at moderate intensity combined with diaphragmatic breathing exercises for 12 weeks, the CON will only attend 3 sessions/week of diaphragmatic breathing exercises for 12 weeks. The lung functions will be assessed by the spirometry testing. The chest expansion will be determined using a tape measurement. Additionally, exercise capacity will be tested using cardiopulmonary exercise testing protocol. All the outcomes will be examined at baseline, and after 12 weeks of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Well controlled fibromyalgia.
* Mild restrictive lung affection.
* Body mass index less than 30kg/m2.
* Moderate level of physical activity.

Exclusion Criteria:

* Any chest diseases.
* Musculoskeletal/ neurological limitations to exercise.
* Smokers.
* Pregnant.

Ages: 30 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2024-11-25 (Estimated); Primary Completion 2025-03-20 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Lung function | At baseline and 12 weeks
  Ventilatory function parameters, including forced vital capacity and forced expiratory volume in the first second will be measured by experienced technicians at baseline and after 12 weeks in all groups using the Medgraphics pulmonary function testing system (Breezesuite Ultima PFX, Milano, Italy) in strict adherence to the guidelines outlined in the user manual.

SECONDARY OUTCOMES:
Chest expansion | At baseline and 12 weeks
  A centimeter tape measure will be used to assess chest expansion, and all measurements will be taken with the patients adopting a straight posture while standing. Two levels of chest expansion will be measured, the axillary level will be evaluated for upper chest expansion assessment, and the xyphoid level will be evaluated for lower chest expansion assessment.
Exercise capacity | At baseline and 12 weeks
  Cardiopulmonary exercise test will be conducted for all women at baseline and post-study based on the guidelines set by the American College of Sports Medicine to determine VO2max for each women.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Sayed Saif, Ph.D, Study Director — National institute for Gerontology

IPD SHARING:
Plan to Share IPD: No